CLINICAL TRIAL: NCT03176134
Title: A Phase III Randomized, Active-comparator-Controlled Clinical Trial to Study the Safety and Efficacy of MK-1986 (Tedizolid Phosphate) and Comparator, in Subjects From Birth to Less Than 12 Years of Age With Acute Bacterial Skin and Skin Structure Infections (ABSSSI)
Brief Title: A Study of Safety and Efficacy of MK-1986 (Tedizolid Phosphate) and Comparator in Participants From Birth to Less Than 12 Years of Age With Acute Bacterial Skin and Skin Structure Infections (MK-1986-018)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1986-018; MK-1986-018 (Other: MSD Protocol Number); 2016-003884-20 (EudraCT Number)
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Acute Bacterial Skin and Skin Structure Infections
MeSH Terms: interventions — tedizolid phosphate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1: Tedizolid phosphate 6 to <12 Years (Experimental): Participants will receive tedizolid phosphate once-daily single 200-mg dose (body weight ≥50 kg) or twice-daily 2-mg/kg doses (body weight 30 kg to <50 kg); or twice-daily 2.5-mg/kg doses (body weight 3.2 kg to <30 kg), by IV and/or oral suspension for 6 to 10 days.
  Interventions: Drug: Tedizolid phosphate
- Cohort 1: Comparator 6 to <12 Years (Active Comparator): Participants will receive comparator IV and/or oral per local standard of care for 10 to 14 days.
  Interventions: Drug: Comparator
- Cohort 2: Tedizolid phosphate 2 to <6 Years (Experimental): Participants will receive tedizolid phosphate once-daily single 200-mg dose (body weight ≥50 kg) or twice-daily 2-mg/kg doses (body weight 30 kg to <50 kg); or twice-daily 2.5-mg/kg doses (body weight 3.2 kg to <30 kg), by IV and/or oral suspension for 6 to 10 days.
  Interventions: Drug: Tedizolid phosphate
- Cohort 2: Comparator 2 to <6 Years (Active Comparator): Participants will receive comparator IV and/or oral per local standard of care for 10 to 14 days.
  Interventions: Drug: Comparator
- Cohort 3: Tedizolid phosphate 28 Days to <2 Years (Experimental): Participants will receive tedizolid phosphate once-daily single 200-mg dose (body weight ≥50 kg) or twice-daily 2-mg/kg doses (body weight 30 kg to <50 kg); or twice-daily 2.5-mg/kg doses (body weight 3.2 kg to <30 kg), by IV and/or oral suspension for 6 to 10 days.
  Interventions: Drug: Tedizolid phosphate
- Cohort 3: Comparator 28 Days to <2 Years (Active Comparator): Participants will receive comparator IV and/or oral per local standard of care for 10 to 14 days.
  Interventions: Drug: Comparator
- Cohort 4: Tedizolid phosphate Birth to <28 Days Term and Preterm Neonates (Experimental): Participants will receive tedizolid phosphate ≤200 mg daily dose, IV and/or oral suspension for 6 to 10 days. Exact mg/kg dose is to be determined based on results of another study (NCT03217565) covering the age range.
  Interventions: Drug: Tedizolid phosphate
- Cohort 4: Comparator Birth to <28 Days Term and Preterm Neonates (Active Comparator): Participants will receive comparator IV and/or oral per local standard of care for 10 to14 days.
  Interventions: Drug: Comparator

INTERVENTIONS:
Drug: Tedizolid phosphate — Tedizolid phosphate IV solution or oral suspension
  Other Names: MK-1986; TR-701 FA
  Arms: Cohort 1: Tedizolid phosphate 6 to <12 Years; Cohort 2: Tedizolid phosphate 2 to <6 Years; Cohort 3: Tedizolid phosphate 28 Days to <2 Years; Cohort 4: Tedizolid phosphate Birth to <28 Days Term and Preterm Neonates
Drug: Comparator — Vancomycin IV, linezolid IV or oral (outside European Union only), clindamycin IV or oral, flucloxacillin IV or oral, cefazolin IV, or cephalexin oral provided locally by the trial site and administered per local standard of care
  Arms: Cohort 1: Comparator 6 to <12 Years; Cohort 2: Comparator 2 to <6 Years; Cohort 3: Comparator 28 Days to <2 Years; Cohort 4: Comparator Birth to <28 Days Term and Preterm Neonates

SUMMARY:
This study will evaluate the safety, tolerability, and efficacy of tedizolid phosphate (MK-1986) compared with comparator antibacterial agent in participants from birth to less than 12 years of age with acute bacterial skin and skin structure infections (ABSSSI).

DETAILED DESCRIPTION:
Participants will be randomized (3:1) to receive tedizolid phosphate at a weight-based dose ≤200 mg/day, intravenous (IV) and/or oral suspension for 6 to 10 days, or comparator IV and/or oral per local standard of care for 10 to 14 days. The switch from IV to oral administration can be made at any time based on 1) no worsening of the primary skin lesion, 2) last temperature <37.7 °C, and 3) primary acute bacterial skin and skin structure infection (ABSSSI) site has not worsened and at least 1 site has improved from Baseline. The potential 4-day treatment extension will be based on clinical need as judged by the investigator, considering the following criteria: 1) ≥40% reduction in primary lesion size, 2) reduction in pain, and 3) no new signs and symptoms and no complications attributable to ABSSSI compared with Baseline.

ELIGIBILITY:
Inclusion Criteria:

* Has a parent/legally acceptable representative who is able to give documented informed consent
* Has acute bacterial skin and skin structure infections (ABSSSI), defined as ≥1 of the following: 1) cellulitis/erysipelas, 2) major cutaneous abscess, or 3) wound infection
* Local symptoms of ABSSSI that started within 14 days before study start
* Suspected or documented Gram-positive bacterial infection

Exclusion Criteria:

* Uncomplicated skin and skin structure infection
* ABSSSI due to or associated with disallowed etiology per protocol
* Received antibacterial therapy for treatment of the current episode of ABSSSI except 1) <48 hours of antibacterial therapy with a short-acting antibacterial drug, or 2) response is considered to be failure (no improvement in signs and symptoms) after at least 48 hours of therapy
* Known bacteremia, severe sepsis, or septic shock
* Significant or life-threatening condition, disease, or organ system condition
* Recent history of opportunistic infections where the underlying cause of the infection is still active, or is suspected to be at risk of opportunistic infection with unusual pathogens
* Received or is receiving treatment for active tuberculosis within 1 month of study start
* Known or suspected severe neutropenia
* Human immunodeficiency virus (HIV) positive and has Cluster of Differentiation (CD) 4 cell count <15% (HIV testing is not required for eligibility)
* Renal impairment that requires renal filtration
* Severe hepatic impairment
* Cardiac or electrocardiogram (ECG) finding that would limit participation in the study
* Received an investigational medicinal product (not approved) within 30 days before study start
* Investigational device present or removed within 30 days before study start
* Previously treated with tedizolid phosphate
* Contraindication, including hypersensitivity to tedizolid phosphate, other oxazolidinones, or any component in the formulation
* Contraindication, including hypersensitivity to all available comparator drugs
* Wound infection and history of hypersensitivity to aztreonam adjunctive therapy or metronidazole adjunctive therapy, if adjunctive therapy is required
* Needs oral administration of methotrexate, topotecan, irinotecan, or rosuvastatin, during administration of oral study drug (administration during the follow-up period, ie, after the end of treatment (EOT) visit, is allowed, as is administration during treatment with IV drug)
* Female who is pregnant or nursing or is of childbearing potential and not abstinent; or male who is not abstinent
* Use of monoamine oxidase inhibitors, tricyclic antidepressants, buspirone, selective serotonin reuptake inhibitors, or serotonin 5-hydroxytryptamine receptor agonists (triptans)
* Identified as having used illicit drugs (urine drug screening not required for entry)

Ages: 1 Day to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (58):
- United States (8):
  - Rady Children's Hospital-San Diego ( Site 0118), San Diego, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago ( Site 0129), Chicago, Illinois
  - Children's Hospital of Michigan ( Site 0100), Detroit, Michigan
  - William Beaumont Hospital ( Site 0108), Royal Oak, Michigan
  - St. Louis Children's Hospital ( Site 0127), St Louis, Missouri
  - Cook Children's Medical Center ( Site 0124), Fort Worth, Texas
  - Baylor College of Medicine - Texas Children's Hospital ( Site 0107), Houston, Texas
  - Children's Hospital of Richmond at VCU ( Site 0123), Richmond, Virginia
- Brazil (4):
  - Hospital Pequeno Principe ( Site 0276), Curitiba, Paraná
  - Inst de Medicina Integral Professor Fernando Figueira- IMIP ( Site 0277), Recife, Pernambuco
  - Centro de Estudos e Pesquisa em Molestias Infecciosas - CPCL-CENTRO DE ESTUDOS E PESQUISAS EM MOLES, Natal, Rio Grande do Norte
  - Instituto D'Or de Pesquisa e Ensino (IDOR)-Hospital São Luiz Jabaquara ( Site 0283), São Paulo
- Bulgaria (9):
  - MHAT Sv. Nikolay Chudotvorets EOOD ( Site 0338), Lom, Montana
  - UMHAT Deva Maria ( Site 0333), Burgas
  - MHAT City Clinic Sv. Georgi EOOD ( Site 0334), Montana
  - MHAT Dr. Stamen Iliev AD ( Site 0339), Montana
  - UMHAT Dr. Georgi Stranski EAD ( Site 0330), Pleven
  - UMHAT Sv. Georgi ( Site 0332), Plovdiv
  - MBAL Medica Ruse EOOD ( Site 0336), Rousse
  - UMHAT Kanev AD ( Site 0337), Rousse
  - UMHATEM. N.I.Pirogov. EAD ( Site 0331), Sofia
- Georgia (4):
  - JSC Evex Hospitals. ( Site 0601), Batumi, Adjara
  - Tbilisi State Medical University G. Zhvania Pediatric Academic Clinic ( Site 0600), Tbilisi, K'alak'i T'bilisi
  - JSC Evex Hospital ( Site 0602), Tbilisi
  - JSC Evex Hospitals ( Site 0603), Tbilisi
- Haunersches Kinderspital ( Site 0480), München, Bavaria, Germany
- Guatemala (3):
  - Clinica Privada ( Site 0551), Guatemala City
  - Private Practice Mario Melgar ( Site 0552), Guatemala City
  - Private Practice Dra. Manrique ( Site 0553), Guatemala City
- Latvia (2):
  - Daugavpils Regional Hospital ( Site 0651), Daugavpils
  - Liepaja Regional Hospital ( Site 0652), Liepāja
- Lithuania (3):
  - Hospital of Lithuanian University of Health Sciences Kaunas ( Site 0701), Kaunas
  - Klaipedos Vaiku Ligonine ( Site 0700), Klaipėda
  - Vaiku ligonine VsI VUL Santaros kliniku filialas ( Site 0702), Vilnius
- Mexico (5):
  - Hospital Civil Fray Antonio Alcalde-pediatrics infectious diseases ( Site 0230), Guadalajara, Jalisco
  - Instituto Nacional de Pediatria ( Site 0231), Mexico City, Mexico City
  - Hospital Infantil de Mexico Federico Gomez ( Site 0227), Mexico City, Mexico City
  - CHRISTUS - LATAM HUB CENTER OF EXCELLENCE AND INNOVATION S.C. ( Site 0241), General Escobedo, Nuevo León
  - Centenario Hospital Miguel Hidalgo-Pediatrics Department ( Site 0239), Aguascalientes
- Poland (3):
  - Wojewodzki Szpital Obserwacyjno Zakazny ( Site 0429), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - SZPZOZ im. Dzieci Warszawy w Dziekanowie Lesnym ( Site 0431), Łomianki, Masovian Voivodeship
  - Wojewodzki Szpital Specjalistyczny im. dr. Wladyslawa Bieganskiego ( Site 0427), Lodz, Łódź Voivodeship
- Russia (3):
  - City Childrens Clinical Emergency Hospital ( Site 0507), Novosibirsk, Novosibirsk Oblast
  - Smolensk Regional Clinical Hospital ( Site 0511), Smolensk, Smolensk Oblast
  - Children s Republican Clinical Hospital ( Site 0512), Kazan', Tatarstan, Respublika
- South Africa (3):
  - Emmed Research Incorporating ( Site 0377), Pretoria, Gauteng
  - Setshaba Research Centre ( Site 0378), Pretoria, Gauteng
  - Enhancing Care Foundation-DICRS ( Site 0381), Durban, KwaZulu-Natal
- Turkey (Türkiye) (7):
  - Cukurova Uni Tip Fak Cocuk Saglıgı ve Hasta ABD ( Site 0353), Adana
  - Hacettepe Universitesi Tip Fakultesi Hastanesi ( Site 0351), Ankara
  - Ankara City Hospital-Infectious Disease and Clinical Microbiology ( Site 0359), Ankara
  - Osmangazi UTF ( Site 0357), Eskişehir
  - Istanbul Universitesi Istanbul Tip Fakultesi ( Site 0355), Istanbul
  - Sisli Hamide Etfal Egitim ve Arastirma Hastanesi ( Site 0358), Istanbul
  - Ege UTF ( Site 0356), Izmir
- Ukraine (3):
  - Dnipropetrovsk Oblast Children's Clinical Hospital ( Site 0868), Dnipro, Dnipropetrovsk Oblast
  - SI Dnipropetrovsk Regional Children Clinical Hospital DOR ( Site 0863), Dnipro, Dnipropetrovsk Oblast
  - Ivano-Frankivsk Regional Children Clinical Hospital ( Site 0865), Ivano-Frankivsk, Ivano-Frankivsk Oblast

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Mngqibisa R, Fofanov O, Grazioso CF, Melgar Toledo M, Boddicker M, Broyde N, Koseoglu S, Romero L, Stevens M, Sears P. A Phase 3 Study of the Safety and Efficacy of Tedizolid Phosphate in Patients <12 Years of Age With Acute Bacterial Skin and Skin Structure Infections. Pediatr Infect Dis J. 2025 Jun 1;44(6):533-538. doi: 10.1097/INF.0000000000004807. Epub 2025 Apr 14. PMID 40233296
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26090&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of100 participants were randomized and received treatment and were evaluable for all safety and efficacy analyses. No participants were enrolled for Cohort 4: Tedizolid phosphate (Birth to <28 Days Neonates) and Cohort 4: Comparator (Birth to <28 Days Term & preterm neonates) arms.
Groups:
- Cohort 1: Tedizolid Phosphate 6 to <12 Years; Cohort 2: Tedizolid Phosphate 2 to <6 Years; Cohort 3: Tedizolid Phosphate 28 Days to <2 Years: Participants received tedizolid phosphate once-daily single 200-mg dose (body weight ≥50 kg) or twice-daily 2-mg/kg doses (body weight ≥30 kg to <50 kg); or twice-daily 2.5-mg/kg doses (body weight 3.2 kg to <30 kg), by IV and/or oral suspension for 6 to 10 days.
- Cohort 1: Comparator 6 to <12 Years; Cohort 2: Comparator 2 to <6 Years; Cohort 3: Comparator 28 Days to <2 Years: Participants received comparator IV and/or oral per local standard of care for 10 to 14 days.
- Cohort 4: Tedizolid Phosphate Birth to <28 Days Term and Preterm Neonates: Participants were to receive Tedizolid phosphate ≤200 mg daily dose, IV and/or oral suspension for 6 to 10 days. Exact mg/kg dose was to be determined based on results of another study (NCT03217565) covering the age range. No participants were enrolled in this arm.
- Cohort 4: Comparator Birth to <28 Days Term and Preterm Neonates: Participants were to receive comparator IV and/or oral as per local standard of care for 10-14 days. No participants were enrolled in this arm.
Period: Overall Study
Arm/Group | Cohort 1: Tedizolid Phosphate 6 to <12 Years | Cohort 1: Comparator 6 to <12 Years | Cohort 2: Tedizolid Phosphate 2 to <6 Years | Cohort 2: Comparator 2 to <6 Years | Cohort 3: Tedizolid Phosphate 28 Days to <2 Years | Cohort 3: Comparator 28 Days to <2 Years | Cohort 4: Tedizolid Phosphate Birth to <28 Days Term and Preterm Neonates | Cohort 4: Comparator Birth to <28 Days Term and Preterm Neonates
Started | 44 | 15 | 16 | 5 | 15 | 5 | 0 | 0
Completed | 42 | 13 | 14 | 5 | 15 | 5 | 0 | 0
Not Completed | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Tedizolid Phosphate 6 to <12 Years | Cohort 1: Comparator 6 to <12 Years | Cohort 2: Tedizolid Phosphate 2 to <6 Years | Cohort 2: Comparator 2 to <6 Years | Cohort 3: Tedizolid Phosphate 28 Days to <2 Years | Cohort 3: Comparator 28 Days to <2 Years | Total
Number analyzed (Participants) | 44 | 15 | 16 | 5 | 15 | 5 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.5 (1.7) | 9.2 (1.4) | 3.1 (1.1) | 3.4 (1.1) | 0.9 (0.2) | 1.0 (0.1) | 6.0 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 8 | 8 | 2 | 11 | 2 | 47
  Male | 28 | 7 | 8 | 3 | 4 | 3 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 5 | 1 | 2 | 1 | 17
  Not Hispanic or Latino | 38 | 13 | 11 | 4 | 13 | 4 | 83
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 9 | 1 | 11
  White | 41 | 15 | 13 | 4 | 4 | 3 | 80
  More than one race | 3 | 0 | 2 | 1 | 1 | 1 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Number of participants who experienced an AE were reported.
Time Frame: Up to approximately 35 days
Population: All randomized participants who received at least one dose of study intervention. No participants were enrolled for Cohort 4: Tedizolid phosphate (Birth to <28 Days Neonates) and Cohort 4: Comparator (Birth to <28 Days Term & preterm neonates) arms. So, cohort 4 arms were not included in the analysis per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Tedizolid Phosphate 6 to <12 Years | Cohort 1: Comparator 6 to <12 Years | Cohort 2: Tedizolid Phosphate 2 to <6 Years | Cohort 2: Comparator 2 to <6 Years | Cohort 3: Tedizolid Phosphate 28 Days to <2 Years | Cohort 3: Comparator 28 Days to <2 Years
Number analyzed (Participants) | 44 | 15 | 16 | 5 | 15 | 5
Participants | 7 | 2 | 7 | 2 | 7 | 2

2. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Number of participants who experienced an AE were reported. The number of participants who discontinued study treatment due to an AE were reported.
Time Frame: Up to approximately day 15
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Tedizolid Phosphate 6 to <12 Years | Cohort 1: Comparator 6 to <12 Years | Cohort 2: Tedizolid Phosphate 2 to <6 Years | Cohort 2: Comparator 2 to <6 Years | Cohort 3: Tedizolid Phosphate 28 Days to <2 Years | Cohort 3: Comparator 28 Days to <2 Years
Number analyzed (Participants) | 44 | 15 | 16 | 5 | 15 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Hematopoietic Cytopenias
Description: Hematopoietic cytopenia is a condition where there is a lower-than-normal amount of one or multiple kinds of blood cells. A standardized Medical Dictionary for Regulatory Activities (MedDRA) query for hematopoietic cytopenia was conducted. The number of participants with a hematopoietic cytopenia were reported.
Time Frame: Up to approximately 35 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Tedizolid Phosphate 6 to <12 Years | Cohort 1: Comparator 6 to <12 Years | Cohort 2: Tedizolid Phosphate 2 to <6 Years | Cohort 2: Comparator 2 to <6 Years | Cohort 3: Tedizolid Phosphate 28 Days to <2 Years | Cohort 3: Comparator 28 Days to <2 Years
Number analyzed (Participants) | 44 | 15 | 16 | 5 | 15 | 5
Participants | 0 | 0 | 1 | 0 | 1 | 0

4. Secondary Outcome: Percentage of Participants With Clinical Response (CR) Per Investigator Assessment
Description: CR was defined as clinical success, failure or indeterminate as per investigator assessment. Success was all of the following: resolution/near resolution of most disease-specific signs & symptoms, absence/near resolution of regional/systemic signs of infection if present at baseline (BL) & no new signs, symptoms, or complications, so, no further antibiotic therapy required. Failure was any of the following: requires additional antibiotic therapy, unplanned major surgical intervention required due to study drug failure, developed osteomyelitis after BL, persistent gram+ bacteremia, treatment emergent adverse event (TEAE) leading to study drug discontinuation & required additional antibiotic therapy to treat infection or death within 28 days of first infusion. Indeterminate was no efficacy data available. Per protocol, percentage of participants with CR for Cohorts 1, 2 & 3 & all cohorts together were reported, & failure & indeterminate responses were pooled.
Time Frame: Up to approximately 25 days
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- All Cohorts: Tedizolid Phosphate: Participants in Cohort 1 (age: 6 to <12 years), Cohort 2 (age: 2 to <6 years), and Cohort 3 (age: 28 days to <2 years) received tedizolid phosphate once-daily single 200-mg dose (body weight ≥50 kg) or twice-daily 2-mg/kg doses (body weight ≥30 kg to <50 kg); or twice-daily 2.5-mg/kg doses (body weight 3.2 kg to <30 kg), by IV and/or oral suspension for 6 to 10 days.
- All Cohorts: Comparator: Participants in Cohort 1 (age: 6 to <12 years), Cohort 2 (age: 2 to <6 years), and Cohort 3 (age: 28 days to <2 years) received comparator IV and/or oral per local standard of care for 10 to 14 days.
Arm/Group | Cohort 1: Tedizolid Phosphate 6 to <12 Years | Cohort 1: Comparator 6 to <12 Years | Cohort 2: Tedizolid Phosphate 2 to <6 Years | Cohort 2: Comparator 2 to <6 Years | Cohort 3: Tedizolid Phosphate 28 Days to <2 Years | Cohort 3: Comparator 28 Days to <2 Years | All Cohorts: Tedizolid Phosphate | All Cohorts: Comparator
Number analyzed (Participants) | 44 | 15 | 16 | 5 | 15 | 5 | 75 | 25
Percentage of Participants
  Clinical Success | 93.2 [81.3 to 98.6] | 86.7 [59.5 to 98.3] | 87.5 [61.7 to 98.4] | 100.00 [47.8 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [47.8 to 100.0] | 93.3 [85.1 to 97.8] | 92.0 [74.0 to 99.0]
  Clinical Failure or Indeterminate | 6.8 [1.4 to 18.7] | 13.3 [1.7 to 40.5] | 12.5 [1.6 to 38.3] | 0.0 [NA to NA] — NA = Lower limit and upper limit of 95%CI were not calculated due to insufficient number of participants with response. | 0.0 [NA to NA] — NA = Lower limit and upper limit of 95%CI were not calculated due to insufficient number of participants with response. | 0.0 [NA to NA] — NA = Lower limit and upper limit of 95%CI were not calculated due to insufficient number of participants with response. | 6.7 [2.2 to 14.9] | 8.0 [1.0 to 26.0]
Statistical Analysis 1: Comparison: Cohort 1: Tedizolid Phosphate 6 to <12 Years vs Cohort 1: Comparator 6 to <12 Years; Test type: Other; Estimated Difference = 6.5, 95% CI 2-sided [-12.2 to 25.3] — The estimated difference in the clinical success rate and 2-sided 95% confidence interval (CI) were calculated using the unstratified method of Miettinen and Nurminen
Statistical Analysis 2: Comparison: Cohort 2: Tedizolid Phosphate 2 to <6 Years vs Cohort 2: Comparator 2 to <6 Years; Test type: Other; Estimated Difference = -12.5, 95% CI 2-sided [-28.7 to 3.7] — The estimated difference in the clinical success rate and 2-sided 95% CI were calculated using the unstratified method of Miettinen and Nurminen
Statistical Analysis 3: Comparison: Cohort 3: Tedizolid Phosphate 28 Days to <2 Years vs Cohort 3: Comparator 28 Days to <2 Years; Test type: Other; Estimated Difference = 0.0, 95% CI 2-sided [0.0 to 0.0] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: All Cohorts: Tedizolid Phosphate vs All Cohorts: Comparator; Test type: Other; Estimated Difference = 1.3, 95% CI 2-sided [-10.7 to 13.4] — [estimate comment as in outcome 4, analysis 2]

5. Secondary Outcome: Percentage of Clinically Evaluable (CE) Participants With CR Per Investigator Assessment
Description: CR was defined as clinical success, failure or indeterminate as per investigator assessment. Success was all of the following: resolution/near resolution of most disease-specific signs & symptoms, absence/near resolution of regional/systemic signs of infection if present at BL & no new signs, symptoms, or complications, so, no further antibiotic therapy required. Failure was any of the following: requires additional antibiotic therapy, unplanned major surgical intervention required due to study drug failure, developed osteomyelitis after BL, persistent gram+ bacteremia, treatment emergent adverse event leading to study drug discontinuation & required additional antibiotic therapy to treat infection or death within 28 days of first infusion. Indeterminate was no efficacy data available. Per protocol, percentage of participants with CR for Cohorts 1, 2 & 3 and all cohorts together were reported, & failure & indeterminate responses were pooled.
Time Frame: Up to approximately 25 days
Population: CE participants included all randomized participants who received at least one dose of study intervention, had a confirmed ABSSSI, had a suspected or documented gram+ infection from BL, received a sufficient course of therapy. No participants were enrolled for Cohort 4: Tedizolid phosphate (Birth to <28 Days Neonates) and Cohort 4: Comparator (Birth to <28 Days Term & preterm neonates) arms. So, cohort 4 arms were not included in the analysis per protocol.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1: Tedizolid Phosphate 6 to <12 Years | Cohort 1: Comparator 6 to <12 Years | Cohort 2: Tedizolid Phosphate 2 to <6 Years | Cohort 2: Comparator 2 to <6 Years | Cohort 3: Tedizolid Phosphate 28 Days to <2 Years | Cohort 3: Comparator 28 Days to <2 Years | All Cohorts: Tedizolid Phosphate | All Cohorts: Comparator
Number analyzed (Participants) | 39 | 13 | 14 | 5 | 15 | 5 | 68 | 23
Percentage of Participants
  Clinical Success | 100.00 [91.0 to 100.0] | 100.0 [75.3 to 100.0] | 100.0 [76.8 to 100.0] | 100.00 [47.8 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [47.8 to 100.0] | 100.00 [94.7 to 100.0] | 100.0 [85.2 to 100.0]
  Clinical Failure or Indeterminate | 0.0 [NA to NA] — NA = Lower limit and upper limit of 95%CI were not calculated due to insufficient number of participants with response. | 0.0 [NA to NA] — NA = Lower limit and upper limit of 95%CI were not calculated due to insufficient number of participants with response. | 0.0 [NA to NA] — NA = Lower limit and upper limit of 95%CI were not calculated due to insufficient number of participants with response. | 0.0 [NA to NA] — NA = Lower limit and upper limit of 95%CI were not calculated due to insufficient number of participants with response. | 0.0 [NA to NA] — NA = Lower limit and upper limit of 95%CI were not calculated due to insufficient number of participants with response. | 0.0 [NA to NA] — NA = Lower limit and upper limit of 95%CI were not calculated due to insufficient number of participants with response. | 0.0 [NA to NA] — NA = Lower limit and upper limit of 95%CI were not calculated due to insufficient number of participants with response. | 0.0 [NA to NA] — NA = Lower limit and upper limit of 95%CI were not calculated due to insufficient number of participants with response.
Statistical Analysis 1: Comparison: Cohort 1: Tedizolid Phosphate 6 to <12 Years vs Cohort 1: Comparator 6 to <12 Years; Test type: Other; Estimated Difference = 0.0, 95% CI 2-sided [0.0 to 0.0] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Cohort 2: Tedizolid Phosphate 2 to <6 Years vs Cohort 2: Comparator 2 to <6 Years; Test type: Other; Estimated Difference = 0.0, 95% CI 2-sided [0.0 to 0.0] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 3: Comparison: Cohort 3: Tedizolid Phosphate 28 Days to <2 Years vs Cohort 3: Comparator 28 Days to <2 Years; Test type: Other; Estimated Difference = 0.0, 95% CI 2-sided [0.0 to 0.0] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 4: Comparison: All Cohorts: Tedizolid Phosphate vs All Cohorts: Comparator; Test type: Other; Estimated Difference = 0.0, 95% CI 2-sided [0.0 to 0.0] — [estimate comment as in outcome 4, analysis 2]

ADVERSE EVENTS:
Time Frame: Up to approximately 35 days
Description: All-cause mortality was reported on all randomized participants. Serious and non-serious AEs were reported on all randomized participants who received at least one dose of study treatment.
Arm/Group | Cohort 1: Tedizolid Phosphate 6 to <12 Years | Cohort 1: Comparator 6 to <12 Years | Cohort 2: Tedizolid Phosphate 2 to <6 Years | Cohort 2: Comparator 2 to <6 Years | Cohort 3: Tedizolid Phosphate 28 Days to <2 Years | Cohort 3: Comparator 28 Days to <2 Years
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/15 | 0/16 | 0/5 | 0/15 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/15 | 0/16 | 0/5 | 0/15 | 0/5
Other Adverse Events (participants affected / at risk) | 4/44 | 2/15 | 7/16 | 2/5 | 7/15 | 2/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Tedizolid Phosphate 6 to <12 Years (N=44) | Cohort 1: Comparator 6 to <12 Years (N=15) | Cohort 2: Tedizolid Phosphate 2 to <6 Years (N=16) | Cohort 2: Comparator 2 to <6 Years (N=5) | Cohort 3: Tedizolid Phosphate 28 Days to <2 Years (N=15) | Cohort 3: Comparator 28 Days to <2 Years (N=5)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Viral diarrhoea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT03176134/Prot_SAP_000.pdf